CLINICAL TRIAL: NCT01713790
Title: Effects of Whole Body Vibration With Stochastic Resonance and Exergames in the Elderly in Need of Care: Effects on Physical Functional Performance
Brief Title: Innovative Training Methods for Frail Elderly in the Training Gain Stage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: Goethe University (Other); Maastricht University Medical Center (Other); Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Heiner Baur (PhD), PhD, Bern University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Main study (PhD)- part II
Record Dates: First submitted 2012-10-14; First posted 2012-10-25 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Poor Performance Status
Keywords: physical functional performance; postural balance; reaction time; mobility; muscle strength; cognition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Training group (Experimental): T0 - Intervention program 3x/ week over 10 weeks: Stochastic resonance whole-body vibration + Exergame + leg press - T1
  Interventions: Device: Stochastic resonance whole-body vibration; Device: Exergame; Device: Leg press

INTERVENTIONS:
Device: Stochastic resonance whole-body vibration — Stochastic resonance whole-body vibration training program over 10 weeks, three times a week with 3 to 6 Hz, Noise 4.
  Other Names: SRT Zeptor® med plus Noise (Swiss Frei AG, Switzerland)
Device: Exergame — training program over 10 weeks, three times a week.
  Other Names: Virtual game board
Device: Leg press — training program over 10 weeks, three times a week.
  Other Names: Swiss Frei AG, Switzerland

SUMMARY:
This study aims to examine long term effects in the training gain stage of the falls management exercise programs (FaME, from Skelton and Dinan) over 10 weeks on physical functional performance after mechanical SR-WBV, dance therapy and strength training intervention in a frail elderly population.

DETAILED DESCRIPTION:
This study is based on the guideline of falls management exercise programs (FaME; from Skelton and Dinan).

The goals:

Skilling up: improvement in neuromuscular control, postural control and strengthening of large muscle groups of the lower extremity.

Training Gain: improvement of functional abilities. Maintaining the Gains: muscle growth, improvement of bone density and multi-sensory exercises.

First, a pilot study was conducted with untrained elderly ("Effects of stochastic resonance therapy on postural control in the elderly population" (KEK Bern: No.228/09, Clinical Trial Registry: NCT01045746). Following, a second pilot study was conducted with frail elderly (Application of Whole-body Vibration With Stochastic Resonance in Frail Elderly: The Effects on Postural Control Clinical Trial Registry: NCT01543243).

It was found that the selected chosen form of recruitment (presentation and advertisement) and the measurements methods are suitable for untrained elderly. But for frail elderly the chosen form of recruitment and the measurement methods are not sufficient.

For this study, adapted measurement parameters for balance, strength and cognition will be used.

The goals of this study:

Evaluate the effects of

* functional lower extremity
* dynamic balance
* reaction time
* mobility
* muscle strength and cognition.

This is a one-group pre-post design study and the participants will be recruited in Canton Bern - Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* RAI (Resident Assessment Instrument) >0
* live in canton Bern
* in terms of training load be resistant.

Exclusion Criteria:

* acut joint disease, acut thrombosis, acute fractures, acute infections, acute tissue damage, or acute -- surgical scars
* seniors with prosthesis.
* alcoholic
* acute joint disease, activated osteoarthritis, rheumatoid arthritis
* acute inflammation or infection tumors
* fresh surgical wounds
* severe migraine
* epilepsy
* acute severe pain

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPBB) | Change from baseline in SPBB at 10 weeks.
  The SPBB assess lower extremity function at baseline and after a 10-week interventions period.

SECONDARY OUTCOMES:
dynamic body balance | Change from baseline in dynamic body balance at 10 weeks.
  The Expanded Timed Get Up-and-Go (ETGUG) will be used for measuring dynamic body balance. At 2, 8 and 10 meters along the walkway, markers were set. In the ETGUG test, times for the component tasks are measured at baseline and after a 10-week interventions period.
walking in single (ST) and dual task (DT) conditions | Change from baseline during walking in ST and DT condition at 10 weeks.
  1. For the single task condition, the participants will be instructed to walk a distance of 20 meters at their self-selected walking speed. Total time were measured.
  2. For the dual task condition, the participant had to count backwards from the number 250 in steps of 7 while walking the same distance at their self-selected walking speed. Total walking times were measured.
     * The time differences between the two tasks are evaluated at baseline and after a 10-week interventions period.
mobility | Change from baseline in mobility at 10 weeks.
  The participants using a StepWatch ™ Activity Monitor (SAM) pedometer. This digital pedometer record the total daily steps at baseline and after a 10-week interventions period.
knee extension maximum voluntary contraction (MVC) | Change from baseline in knee extension MVC at 10 weeks.
  It will be evaluated by isometric MVC at 90 degree angle in the knee joint at baseline and after a 10-week interventions period.
knee extension rate of force develompent (RFD) | Change from baseline in knee extension RFD at 10 weeks.
  It will be evaluated by isometric RFD at 90 degree angle in the knee joint at baseline and after a 10-week interventions period.
knee flexion maximum voluntary contraction (MVC) | Change from baseline in knee flexion MVC at 10 weeks.
  It will be evaluated by isometric MVC at 90 degree angle in the knee joint at baseline and after a 10-week interventions period.
knee flexion rate of force develompent (RFD) | Change from baseline in knee flexion RFD at 10 weeks.
  It will be evaluated by isometric RFD at 90 degree angle in the knee joint at baseline and after a 10-week interventions period.

CONTACTS AND LOCATIONS:
Overall Officials: Slavko Rogan, MSc, Study Chair — Bern University of Applied Science, Department WGS; Lorenz Radlinger, PhD, Study Director — Bern University of Applied Science, Department WGS; Dietmar Schmidtbleicher, Prof., PhD, Study Director — Johann Wolfgang Goethe University, Department Sport Science; Rob de Bie, Prof., PhD, Study Director — University Maastricht, Department Epidemiology; Eling D de Bruin, Prof., PhD, Study Director — Swiss Federal Institute of Technology Zurich, Department Human Movement Science; Baur Heiner, PhD, Principal Investigator — Bern University of Applied Sciences
Locations (1):
- Slavko Rogan, Bern, Canton of Bern, Switzerland